CLINICAL TRIAL: NCT04541966
Title: What Happens to First Trimester Nuchal Translucency Greater Than or Equal 99ème Percentile and Inferior 3.5 mm
Brief Title: What Happens to First Trimester Nuchal Translucency
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0479
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-06

CONDITIONS: Nuchal Translucency
Keywords: Ultrasound abnormalities; Genetic abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nuchal translucency> = 99th percentile and <3.5mm: Nuchal translucency> = 99th percentile and <3.5mm
- Nuchal translucency> = 3.5 mm: Nuchal translucency> = 3.5 mm

SUMMARY:
First trimester nuchal translucency is a call point for genetic abnormalities and birth defects. Nuchal translucency varies with LCC and therefore with gestational age as described by Chung et al who created a 99th percentile curve of nuchal translucency versus LCC. The majority of centers use the 3.5 mm cutoff as the 99th percentile instead of using nuchal translucency based on LCC. The objective of this study is to compare the fate of nuchal hyperclites> = 99th p but <3.5mm versus 3.5mm. For this the investigators have studied the ultrasound and genetic abnormalities. The investigators were also interested in the pregnancy outcomes and the percentage of pregnancies in the group> = 99th p and <3.5mm that would have been sampled for a high combined risk for trisomy 21, and therefore to determine the benefit of a systematic sample. for HCN as well as the interest of performing an ACPA that would not be performed on a sample with a high risk of trisomy 21.

ELIGIBILITY:
Inclusion criteria:

nuchal translucency> = 99th percentile

Exclusion criteria:

- multiple pregnancies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Single pregnancies with nuchal hyperclarity in the first trimester> = 99th percentile at the Montpellier University Hospital with early pregnancy between January 2017 and December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Pregnancies without ultrasound or genetic abnormalities | immediate antenatal and postnatal period
  Pregnancies without ultrasound or genetic abnormalities

SECONDARY OUTCOMES:
ACPA interest | immediate antenatal and postnatal period
  ACPA interest
percentage of samples for high risk combined for trisomy 21 | immediate antenatal and postnatal period
  percentage of samples for high risk combined for trisomy 21
Pregnancy outcomes | immediate antenatal and postnatal period
  Pregnancy outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Florent FUCHS, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC